CLINICAL TRIAL: NCT00563082
Title: Prothrombin Gene Varitaion and Risk of SLE and CHD
Brief Title: Analyzing the Association of Gene Variants With Increased Risk of Coronary Heart Disease in Women With Systemic Lupus Erythematosus
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1393; R01HL088648 (NIH); R01HL088648-01 (NIH)
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2014-03

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: SLE; Genetics
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA and serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: SLE participants positive for both APA and CHD
- 2: Normal participants with a high titer of APA

SUMMARY:
Systemic lupus erythematosus (SLE) is an autoimmune disease that predominantly affects younger premenopausal women. The risk of coronary heat disease (CHD) in women with SLE is up to 50 times higher than in the general population. The conventional risk factors are insufficient to explain this increased risk of CHD in SLE-affected women. This study will perform genetic analysis to determine if genetic variation in the F2 gene is associated with both SLE risk and CHD risk in women with SLE.

DETAILED DESCRIPTION:
SLE is a condition of chronic inflammation of the internal organs, caused by an autoimmune disease. An autoimmune disease is a disorder in which the body's immune system attacks its own tissues through production of abnormal antibodies in the blood. Current treatments for SLE focus on reducing inflammation and production of unusual antibodies. While the exact cause of SLE is unknown, genetics, drugs, viruses, and ultraviolent light are all possible contributors. Previous genetic studies have determined that antiphospholipid antibodies (APA) are present in 50% of people with SLE compared with only 1 to 5% in the general U.S. white population. These antibodies interfere with standard blood vessel function, resulting in blood clots and narrowing of vessels. The F2 gene codes for prothrombin, a precursor of thrombin, which is a key enzyme in blood clotting. Prothrombin can be detected by APA as an antigen, resulting in anti-F2 antibodies. Recent studies have reported the association of F2 genetic variants with non-fatal heart attack, further suggesting that the F2 gene and APA play a role in CHD. In addition to being a biological candidate gene for CHD, F2 is also a positional candidate gene for SLE, as it is close to a region of linkage for SLE on chromosome 11. This study will perform genetic analysis to determine if genetic variation in the F2 gene is associated with both SLE risk and CHD risk in women with SLE.

Using genetic analysis techniques, this study will examine previously collected case-control samples of serum DNA. Study researchers will resequence the entire F2 gene and then examine the role of sequence variations in relation to SLE and the risk of CHD in SLE patients. Researchers will identify rare and common variants of the F2 gene and further screen variants to determine gene-trait relations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLE

Exclusion Criteria:

* Pregnant

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include genetic samples from women with SLE and CHD and from normal control women. The population will be 80.5% U.S. white women and 19.5% U.S. black women.
Sampling Method: Non-Probability Sample
Enrollment: 1254 (Actual)
Dates: Start 2000-05; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Rare and common variants of F2 that contribute to SLE risk and CHD risk in SLE | Measured at Year 4

CONTACTS AND LOCATIONS:
Overall Officials: M. Ilyas Kamboh, PhD, Principal Investigator — University of Pittsburgh